CLINICAL TRIAL: NCT07164924
Title: Evaluation of the Impact of Multiple Sclerosis and Its Treatments on Women Fertility
Acronym: FERTIMUS
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Observatoire Français de la sclérose en plaques (OFSEP) (Unknown); Roche Diagnostic Ltd. (Industry); ARSEP foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2024-CF243
Record Dates: First submitted 2025-03-06; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2024-07

CONDITIONS: Multiple Sclerosis; Neuromyelitis Optica Spectrum Disorders; Fertility
Keywords: Fertility; Anti-Mullerian Hormone (AMH); Multiple sclerosis (MS); Female; Disease activity
MeSH Terms: conditions — Multiple Sclerosis; Neuromyelitis Optica

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — serum for antimüllerian l(AMH) level
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- MS / NMOSD female patients: MS / NMOSD female patients , aged between 18 and 35, with or without MS treatment
  Interventions: Biological: blood sample to analyse AMH level on the serum

INTERVENTIONS:
Biological: blood sample to analyse AMH level on the serum — Evaluation of MS/NMOSD inflammatory activity on the serum AMH level (ng/ml)

SUMMARY:
CONTEXT A desire for pregnancy is common in young patients with multiple sclerosis (MS). The impact of MS on women fertility is debated, and the impact of disease-modifying therapies (DMTs) on fertility is not well known. Antimüllerian hormone (AMH) is a representative biomarker of ovarian reserve that can be used to explore this issue.

OBJECTIVES To examine the impact of MS activity and related DMTs on ovarian reserve measured by serum AMH level.

METHODOLOGY Retrospective multicentre study based on clinical and blood samples from patients included in the OFSEP cohort. A serum sample from more than 800 MS and 96 NMOSD women aged 18-35 will be available for AMH dosing. The results obtained will be interpreted taking into account the age, the inflammatory activity of the disease, the disability (EDSS) and the previous and current DMTs used.

STATISTICAL ANALYSIS Spearman correlation coefficient will be calculated in univariate analysis between serum AMH level and number of relapses that occurred during the 2 years before blood sample collection. For multivariable analysis, multiple mixed linear regression will be performed with AMH level as dependant outcome and number of relapses, age, DMTs (highly active, moderately active or no treatment), disease duration and disability (measured using EDSS) as independent variables. The center will be considered as random-effect. For AMH level categorized as normal or not, mixed logistic regression will be performed with aforementioned covariates. These analyses will be completed by a mediation analysis between AMH level, number of relapses and DMTs with age, EDSS and disease duration as adjustments covariates.

EXPECTED RESULTS :

Evaluation of the potential relationship between AMH levels and MS or NMOSD activity at the first years of the illness.

Evaluation of the potential impact of MS and NMOSD treatments on ovarian reserve.

Optimization of the indications of fertility preservation for MS and NMOSD female patients.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Diagnosis of MS (including CIS) or NMOSD
* Aged 18 to 35 years old at blood sample collection

Exclusion Criteria:

* Diagnosis of radiologically isolated syndrome (RIS)
* Age less than18 or more than 35.
* History of ovarian surgery
* Endometriosis
* Hypergonadotropin amenohrrea
* Any associated known autoimmune disease other than MS
* Previous MS treatment with immunosuppressive agents such as azathioprine, cyclophosphamide, mitoxantrone, bone marrow transplantation
* Previous treatment with gonadotoxic drugs (eg chemotherapy)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women, with age between 18 at 35, with a diagnosis of MS or NMOSD , present in EDMUS database, which has a blood sample in the OFSEP cohort
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2024-12-08 (Actual); Study Completion 2024-12-08 (Actual)

PRIMARY OUTCOMES:
the evaluation of MS/NMOSD inflammatory activity on the serum AMH level (ng/ml) | period of 2 years before blood samples
  Disease activity will be evaluated on the number of relapses that occurred during the 2 years before blood sample collection and total number of relapses, taking disease duration into account.
  The measurement of AMH level will be performed using the electrochemiluminescence method with a Cobas® e411 analyzer (Roche Diagnostics, Meylan, France). This immunoassay is based on a sandwich format between the analyte and the two antibodies: a biotinylated AMH-specific mouse monoclonal capture antibody and a second ruthenium-labeled AMH mouse monoclonal antibody. This assay is a fully automated, robust and precise method. Repeatability and intermediate precision calculated on serum samples range from 1.1% to 1.8% and 3.3% to 4.4%, respectively. The assay time is 18 minutes and the measuring range is from 0.01 to 23 ng/ml. The threshold of inf at1 ng/ml will be considered to be a proof of severe decrease in ovarian reserve

SECONDARY OUTCOMES:
Evaluation of the potential impact of previous treatments used on AMH level | period before the collection of AMH level
  The treatments used will be pooled in highly active treatments (NATALIZUMAB, FINGOLIMOD, PONESIMOD, OFATUMUMAB, ALEMTUZUMAB, CLADRIBINE, OCRELIZUMAB, RITUXIMAB), moderately active (INTERFERON BETA, ACETATE DE GLATIRAMERE, DIMETHYLFUMARATE, LAQUINIMOD, MYCOPHENOLATE MOFETIL, METHOTREXATE) or no treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Clavelou, Principal Investigator — CHU de Clermont-Ferrand
Locations (27):
- France (26):
  - CHU Amiens, Amiens
  - CHU Besancon, Besançon
  - CHU Bordeaux, Bordeaux
  - CHU Caen, Caen
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - AP-HP - Créteil, Créteil
  - CHU Dijon, Dijon
  - CHU Grenoble, Grenoble
  - CHU Lille, Lille
  - CHU Limoges, Limoges
  - Hospices Civils de Lyon, Lyon
  - AP-HM, Marseille
  - CHU Montpellier, Montpellier
  - CHU Nancy, Nancy
  - CHU Nantes, Nantes
  - CHU Nice, Nice
  - CHU Nîmes, Nîmes
  - Hôpital de la Pitié-Salpêtrière, Paris
  - Hôpital Fondation Rothschild, Paris
  - Hôpital Saint Antoine, Paris
  - CHI Poissy- Saint-Germain-en-Laye, Poissy
  - CHU Poitiers, Poitiers
  - CHU Rennes, Rennes
  - CHU Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse
  - CHU Tours, Tours
- CHU Fort-de-France, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: No